CLINICAL TRIAL: NCT05464485
Title: Anterior Cruciate Ligament Hamstring Study: Hamstring Muscle Strength After Anteromedial Portal ACL Reconstruction Versus Tape Locking Screw ACL Reconstruction
Brief Title: Hamstring Muscle Strength After ACL Hamstring Reconstruction
Acronym: HAMSTRING
Status: Completed | Type: Observational
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Bart Robben, MD, Isala
Other Study IDs: 60029.075.16
Record Dates: First submitted 2022-07-10; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACL hamstring reconstructions using semitendinosus (ST) tendon only
  Interventions: Procedure: ACL hamstring reconstructions using semitendinosus (ST) tendon only
- ACL hamstring reconstructions using semitendinosus and gracilis (ST/G) tendon
  Interventions: Procedure: ACL hamstring reconstructions using semitendinosus and gracilis (ST/G) tendon

INTERVENTIONS:
Procedure: ACL hamstring reconstructions using semitendinosus (ST) tendon only — ACL reconstruction with a ST tendon graft received a reconstruction according to the Tape Locking Screw technique (FH Industrie, Quimper, France) with a dedicated interference screw
  Groups: ACL hamstring reconstructions using semitendinosus (ST) tendon only
Procedure: ACL hamstring reconstructions using semitendinosus and gracilis (ST/G) tendon — ACL reconstruction with a ST/G tendon graft received a reconstruction with the anteromedial portal technique with endobutton fixation (Smith & Nephew, London, UK).
  Groups: ACL hamstring reconstructions using semitendinosus and gracilis (ST/G) tendon

SUMMARY:
Anterior Cruciate Ligament (ACL) reconstructions using hamstring grafts can be performed using one or two hamstring grafts, the semitendinosus (ST) tendon only, or both the semitendinosus and gracilis (ST/G) tendon. As most patients strive to return to sport nine months after reconstruction the purpose of this study was to compare the recovery of hamstring muscle strength during these first nine months after reconstruction using the ST or ST/G tendons.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) reconstruction techniques are developing continuously. Studies have shown that anatomical positioning of the femur tunnel is an important predictor for the clinical outcome. This has led to the development of new reconstruction techniques with a more anatomical placement of the femur tunnel: the anteromedial portal (AMP) ACL reconstruction technique and, more recently, the tape locking screw (TLS) ACL reconstruction technique. Multiple retrospective studies have shown that patients have a better short term clinical outcome when the anteromedial portal (AMP) or the tape locking crew (TLS) reconstruction technique is used. At this moment, the most widely used technique is the AMP (performed in approximately 80% of the ACL reconstructions). The TLS technique is widely used in France and the available literature shows good short-term results.

A difference between the AMP and the TLS technique is that the AMP technique uses a double-bundle hamstring graft where the TLS technique uses a single-bundle hamstring graft. The idea is that using a single-bundle hamstring graft causes less hamstring muscle strength deficit. The available literature shows different outcomes of hamstring muscle strength deficit, although, there are no studies found in which the difference in hamstring muscle strength deficit between both techniques directly has been investigated.

Objective: The main objective of this study is to compare the hamstring muscle strength deficit after AMP and TLS reconstruction techniques.

The primary aim of this study is to investigate if there is a difference in hamstring muscle strength deficit at 60°/s flexion in patients with an ACL rupture (18-60 years) who received a tape locking screw ACL reconstruction versus patients who received an anteromedial portal ACL reconstruction 12 weeks after surgery.

The secondary aim of this study is to investigate if there is a difference in muscle strength deficit at 180°/s and 240°/s flexion and extension 12 weeks after surgery and 60°/s, 180°/s and 240°/s flexion and extension 20 weeks after surgery in patients who received a tape locking screw ACL reconstruction versus patients who received an anteromedial portal ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years and younger than 60 years old.
* Mentally competent to understand the informed consent.
* Patient underwent AMP or TLS ACL reconstruction surgery or will undergo AMP or TLS ACL reconstruction surgery

Exclusion Criteria:

* ACL reconstruction surgery older than 12 weeks.
* Meniscus rupture larger than 25%
* Indication for meniscal repair.
* Injury of the collateral ligaments or posterior cruciate ligament
* History of ACL or meniscal rupture
* Neurological or systemic disorder that inhibit adequate rehabilitation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the Orthopaedic outpatient clinic of the Isala in Zwolle if the patient has an ACL rupture and if there is an indication for surgical reconstruction with the AMP or TLS ACL reconstruction technique or at the (standard) 6 weeks follow-up appointment after AMP or TLS ACL reconstruction surgery
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Isokinetic muscle strength deficit | 38 weeks post-surgery
  Comparing isokinetic muscle strength deficit (measured at 60°/s, 180°/s and 240°/s flexion with a the Biodex dynamometer) between both groups

SECONDARY OUTCOMES:
Change in isokinetic muscle strength deficit | 12, 20 and 38 weeks post-surgery
  Comparing the change in isokinetic muscle strength deficit (measured at 60°/s, 180°/s and 240°/s flexion with a the Biodex dynamometer) at 12, 20 and 38 weeks post-surgery

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due institutional privacy guideline but are available from the corresponding author on reasonable request